CLINICAL TRIAL: NCT02299076
Title: Software to Translate Behavioral Economics Insights to Improve Health (Phase 2b)
Brief Title: Pro-Change Smoking Cessation Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VAL Health, LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Rhode Island Primary Care Physicians Corporation (Unknown); Pro-Change Behavior Systems (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R44AG044872-03 (NIH); 5R44AG044872-03 (NIH)
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Smoking Cessation; Motivation
Keywords: Tobacco smoking cessation; Motivation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care with minimal incentives (Other): Participants in this arm receive usual care from the Pro-Change smoking cessation program, and receive compensation for enrolling and completing a survey at the end of the study.
  Interventions: Other: Minimal incentives
- Usual care with BE incentives (Active Comparator): Participants in this arm receive usual care from the Pro-Change smoking cessation program, the chance to win money based on their behavior (behavioral economics incentives), and receive compensation for enrolling and completing a survey at the end of the study.
  Interventions: Behavioral: Behavioral economics incentives

INTERVENTIONS:
Behavioral: Behavioral economics incentives — Behavioral economics-informed incentives to promote engagement and outcomes in a smoking cessation intervention.
  Arms: Usual care with BE incentives
Other: Minimal incentives — Minimal financial incentives to promote engagement and outcomes in a smoking cessation intervention.
  Arms: Usual care with minimal incentives

SUMMARY:
The purpose of this study is to determine whether a behavioral economics solution impacts smoking cessation program engagement and quit rates.

DETAILED DESCRIPTION:
The behavioral economics solution is a weekly regret contest in which participants can win or miss out on money based on their behavior.

ELIGIBILITY:
Inclusion Criteria:

* Be current tobacco users (specifically smokers)
* Be 18 years old or over

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Horgan, MBA, Principal Investigator — President; Kevin Volpp, MD, PhD, Study Director — Scientific Advisory Board; David Asch, MD, Study Director — Scientific Advisory Board
Locations (1):
- VAL Health, Old Greenwich, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January to March, 2016. Recruitment methods: Physician and nurse referrals from Rhode Island Primary Care Physicians Corporation and Facebook advertisements.
  Intake method: Digital intake form hosted by Pro-Change.
Pre-assignment Details: We identified and discontinued 34 participants whose accounts were were flagged as being suspicious. Duplicate accounts were erroneously created by a participant and thus were removed from the study. Suspicious accounts contained personal information identical to existing participants and after investigation, were concluded to be fraudulent.
Groups:
- Usual Care With Minimal Incentives: Participants in this arm receive usual care from the Pro-Change smoking cessation program, and receive compensation for enrolling and completing a survey at the end of the study.
  Minimal incentives: Minimal financial incentives to promote engagement, and outcomes in a smoking cessation intervention.
Period: Overall Study
Arm/Group | Usual Care With Minimal Incentives | Usual Care With BE Incentives
Started | 230 | 226
Completed | 210 | 212
Not Completed | 20 | 14
Not completed — Fraudulent Entries | 20 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care With Minimal Incentives | Usual Care With BE Incentives | Total
Number analyzed (Participants) | 210 | 212 | 422
Age, Continuous [Mean (Full Range); unit: years] | 44 [20 to 79] | 44 [20 to 74] | 44 [20 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 150 | 288
  Male | 72 | 62 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 18 | 27
  Not Hispanic or Latino | 196 | 188 | 384
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 210 | 212 | 422

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Completed Sessions Per Participant
Description: Engagement rates for the intervention will be higher relative to the control arm. Engagement is measured by the number of complete tobacco cessation sessions per participant.
Time Frame: Every 30 days for up to 6 months post-enrollment
Measure: Mean (Inter-Quartile Range); unit: Average Number of Sessions
Units Other Than Participants: Sessions
Arm/Group | Usual Care With Minimal Incentives | Usual Care With BE Incentives
Number analyzed (Participants) | 210 | 212
Number analyzed (Sessions) | 343 | 647
Average Number of Sessions | 1.633 [1 to 2] | 3.052 [1 to 5]
Statistical Analysis 1: Comparison: Usual Care With Minimal Incentives vs Usual Care With BE Incentives; Test type: Superiority — Welch Two Sample t-test; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Outcome of Smoking Cessation Intervention
Description: Quit levels for the intervention will be higher relative to the control arm. Quit level is defined as a participant who progresses to the stage in the tobacco cessation program where they quit smoking. The quit stages are levels 4 and 5 of the tobacco cessation program.
Time Frame: Every 30 days for up to 6 months post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care With Minimal Incentives | Usual Care With BE Incentives
Number analyzed (Participants) | 210 | 212
Participants | 38 | 63

ADVERSE EVENTS:
Time Frame: Up to 6 months post-enrollment.
Description: No adverse events reported.
Arm/Group | Usual Care With Minimal Incentives | Usual Care With BE Incentives
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/212
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/212
Other Adverse Events (participants affected / at risk) | 0/210 | 0/212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes